CLINICAL TRIAL: NCT02095782
Title: Intercalated Combination of Chemotherapy and Erlotinib in 1st Line Setting for Patients Advanced Stage Non-small-cell Lung Cancer With Low Abundant Activating EGFR Mutation(INNOVATE)
Brief Title: Chemotherapy and Erlotinib for Lung Cancer With Low Abundance Epidermal Growth Factor Receptor Mutation
Acronym: INNOVATE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Because of the very slow enrollment, this study was stopped.
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Principal Investigator, Yi-Long Wu, Dr., Guangdong Association of Clinical Trials
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTONG1307
Record Dates: First submitted 2014-03-19; First posted 2014-03-26 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Non-small-cell Lung Cancer
Keywords: non-small cell lung cancer; erlotinib; chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- chemotherapy and erlotinib (Experimental): Intercalated combination of chemotherapy and erlotinib in 1st line setting for patients with advanced stage non-small-cell lung cancer with low abundant activating EGFR mutation
  Interventions: Drug: Intercalated combination of chemotherapy and erlotinib

INTERVENTIONS:
Drug: Intercalated combination of chemotherapy and erlotinib — Primary therapy stage:
  Paclitaxel Patients receive six cycles of Paclitaxel (175 mg/m² on days 1 of a 4 week cycle, intravenously) plus carboplatin (AUC=5, intravenously on day 1 of a 4 week cycle, intravenously) with sequential erlotinib (150 mg/day) on days 8-21 of each cycle.
  Maintenance therapy stage:
  Patients, who complete 6 cycles of therapy without progression or intolerable toxicity, receive erlotinib (150 mg/day) as maintenance therapy until progression, intolerable toxicity or death.
  Other Names: paclitaxel plus carboplatin and targeted therapy erlotinib

SUMMARY:
This is a single arm phase II clinical trial, which aims to evaluate the effectiveness of intercalated combination of doublet chemotherapy of paclitaxel plus carboplatin and erlotinib on patients with advanced stage non-small-cell lung cancer with low abundant activating EGFR mutation.

DETAILED DESCRIPTION:
Primary therapy stage:

Paclitaxel Patients receive six cycles of Paclitaxel (175 mg/m² on days 1 of a 4 week cycle, intravenously) plus carboplatin (AUC=5, intravenously on day 1 of a 4 week cycle, intravenously) with sequential erlotinib (150 mg/day) on days 8-21 of each cycle.

Maintenance therapy stage:

Patients, who complete 6 cycles of therapy without progression or intolerable toxicity, receive erlotinib (150 mg/day) as maintenance therapy until progression, intolerable toxicity or death.

ELIGIBILITY:
Inclusion Criteria:Patients with histologically documented, locally advanced or recurrent (stage IIIb and not amenable to combined modality treatment) or metastatic (stage IV) non-small cell lung cancer.

Low abundant activating EGFR mutation: EGFR exon 19 deletion or exon 21 L858R, which are positive by real-time PCR methods and negative by standard sequencing methods.

Uncommon EGFR mutations are included excluding exon 20 mutations. ECOG performance status of ≤ 2. Patients can administer first line setting of platinum based chemotherapy. Patients must have measurable disease according to the RECIST (version 1.1) criteria.

* Life expectancy of at least 12 weeks.
* Age ≥ 18 years.
* Written (signed) informed Consent to participate in the study.
* Adequate organ function as defined by the following criteria:

Liver function: SGOT (AST) and SGPT (ALT) ≤ 2.5 X ULN in the absence of liver metastases or up to 5 X ULN in case of liver metastases. Total bilirubin ≤ 1.5ULN.

Bone marrow function: Granulocyte count ≥ 1,500/mm3 and platelet count ≥100,000/mm3 and hemoglobin ≥90g/dl.

Renal function: serum creatinine ≤ 1.5 ULN or creatinine clearance ≥ 60 ml/min. (based on modified Cockcroft-Gault formula).

* For all females of childbearing potential a negative serum/urine pregnancy test must be obtained within 48 hours before enrollment. Postmenopausal women must have been amenorrhoeic for at least 12 months to be considered of non-childbearing potential.

Exclusion Criteria:Patients with prior chemotherapy or systemic anti-cancer therapy including target therapy targeting HER family members (such as erlotinib, gefitinib, cetuximab, trastuzumab, etc). Previous adjuvant or neo-adjuvant treatment for non-metastatic disease is permitted if completed ≥ 6 months before the enrollments.

* Patients with history of any other malignancies within 5 years (except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer).
* Patients who have brain metastasis or spinal cord compression. It is permitted if the patient has been treated with surgery and/or radiation with evidence of stable disease for at least 4 weeks.
* Patients who are at risk (in the investigator's opinion) of transmitting human immunodeficiency virus (HIV) through blood or other body fluids.
* Nursing or lactating women.
* Sexually active males and females (of childbearing potential) unwilling to practice contraception during the study.
* Unwilling to write informed consent to participate in the study.
* Patients who is unwilling to accept the follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-03; Primary Completion 2017-01-20 (Actual); Study Completion 2017-01-20 (Actual)

PRIMARY OUTCOMES:
Progression free survival defined by imagery methods | 8 weeks
  From start of anti-cancer therapy untill progression or death

SECONDARY OUTCOMES:
Toxicities related to anti-cancer therapy | 8 weeks
  From start of anti-cancer therapy till progression of death

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Long Wu, Study Chair — Guangdong General Hospital (GGH)& Guangdong Academy of Medical Sciences; Zhen Wang, PhD, Principal Investigator — Guangdong General Hospital & Guangdong Academy of Medical Sciences
Locations (1):
- Guangdong General Hospital & Guangdong Academy of Medical Sciences, Guangzhou, Guangdong, China